CLINICAL TRIAL: NCT04316975
Title: Utility Of Mutational Load As A Predictor For Endoscopic Treatment Response In Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Interpace Diagnostics Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-0679
Record Dates: First submitted 2020-02-24; First posted 2020-03-20 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Barretts Esophagus With Dysplasia; Intramucosal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Subjects will undergo a standard of care (SOC) esophagogastroduodenoscopy (EGD). At this visit, research biopsies will be obtained - 4 research biopsies at the midpoint of current Barrett's Esophagus (BE) OR slides will be cut from clinical Endoscopic Mucosal Resection (EMR). Slides will be analyzed for mutational load (ML) analysis and gastroenterologist (GI) pathologist diagnosis for the presence of adenocarcinoma or degrees of dysplasia. ML will be correlated to the pathology diagnosis on this research biopsy. Subjects will then undergo (Endoscopic Eradication Therapy) EET per routine standard of care at the treating institution until Complete Eradication of Intestinal Metaplasia (CEIM) is achieved. Subjects will be followed (data collection only) during treatment period until CEIM is achieved. After subjects reach CEIM, four additional research biopsies will be collected, from the midpoint of previous BE site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy: Barrett's Esophagus, Intramucosal adenocarcinoma (Other): Subjects will undergo standard of care (SOC) standard esophagogastroduodenoscopy (EGD) for the treatment of their condition (BE or IMC). Four (4) research biopsies will be taken from the midpoint of current disease. In cases where EMR (Endoscopic Mucosal Resection) is performed clinically, no research biopsies will be taken. Following CEIM, four (4) additional research biopsies will be collected, from the midpoint of previous BE site.
  Laboratory Biomarker Analysis: Correlative studies
  Esophagogastroduodenoscopy: Standard of care, research biopsies will be collected if clinical biopsies are taken
  Interventions: Other: Study Driven Procurement of Biopsies

INTERVENTIONS:
Other: Study Driven Procurement of Biopsies — Four research biopsies collected at the midpoint of current BE or IMC at Baseline and after reaching CEIM. Biopsies will be used to calculate ML scores both pre and post EET.
  Other Names: Research Biopsies

SUMMARY:
To evaluate association between mutational load (ML) from esophageal biopsy specimens in pre-endoscopic eradication therapy (EET) in Barrett's Esophagus (BE) or Intramucosal adenocarcinoma (IMC) patients and treatment resistance (treatment resistance will be defined as disease recurrence and/or need for additional intervention such as increased acid suppression, need for anti-reflux surgery, or use of alternate ablative modality).

DETAILED DESCRIPTION:
Potential subjects will be identified via protocol and Institutional Review Board (IRB) methods prior to obtaining written informed consent. Once written informed consent is obtained, subjects will continue with planned routine care upper endoscopy. During the first study visit an upper endoscopy will be performed. At this visit, research specimens will be obtained for mutational load (ML) analysis and gastroenterologist (GI) pathologist diagnosis for the presence of adenocarcinoma or degrees of dysplasia. ML will be correlated to the pathology diagnosis on this research biopsy. Subjects will then undergo EET per routine standard of care at the treating institution until CEIM achieved. Subjects will be followed (data collection only) during treatment period until CEIM is achieved. After subjects reach CEIM, four additional research biopsies will be collected, from the midpoint of previous BE site.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of endoscopic treatment therapy for BE
* Previously untreated "treatment naïve" disease history with confirmed histopathology analysis of at least one of the following:

  * Low- or high-grade dysplastic BE (history of endoscopic mucosal resection (EMR)) is allowable or
  * Intramucosal adenocarcinoma (IMC)
* BE lesion length of at least: C0, M1
* At least 18 years of age at time of consent
* Able and willing to provide written informed consent
* Able and willing to comply with required study procedures and follow-up schedule

Exclusion Criteria:

* History of endoscopic intervention for the treatment of gastroesophageal reflux disease (GERD), BE, or IMC (prior EMR is allowable)
* Current esophageal stenosis/stricture preventing advancement of a therapeutic scope or significant esophageal anatomic abnormalities (masses, obstructive lesions, etc.)
* Dysplasia of intestinal metaplasia (IM) confined only to the gastric cardia (BE Prague Criteria: C0M0)
* Uncontrolled coagulopathy
* Severe medical comorbidities precluding endoscopy, or limiting life expectancy to less than 2 years in the judgment of the endoscopist
* Known portal hypertension, visible esophageal varices, or history of esophageal varices
* Previous esophagectomy surgery involving the gastroesophageal junction (history of a fundoplication is OK)
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation
* Subject has any condition that, in the opinion of the investigator or sponsor, would interfere with accurate interpretation of the study endpoints or preclude participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Correlation of Mean Mutational Load (ML) and Treatment Resistance | Baseline until Month 24
  Treatment resistance will be assessed as a dichotomous variable and defined as those with one or more of the following features: disease recurrence, need for increased acid suppression, need for anti-reflux surgery, or use of alternate ablative modality. The association between pre-EET ML and treatment resistance will be calculated using the difference between the two mean ML values.

SECONDARY OUTCOMES:
Correlation of Mutational Load and Dysplasia Category | Day 1, at enrollment
  The worst pathologic diagnosis at baseline will be recorded and ML between the three dysplasia groups (low grade dysplasia, high grade dysplasia, and esophageal adenocarcinoma) will be compared.
Correlation of Mutational Load and Number of Ablation Sessions to CEIM | From Baseline until the date of first documentation of CEIM, assessed up to 24 Months
  ML calculation will be compared to number of sessions required to achieve CEIM.
Correlation of Mutational Load and Stricture Formation | From Baseline until the date of first documentation of CEIM, assessed up to 24 Months
  ML calculation will be compared to stricture rates.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No